CLINICAL TRIAL: NCT07116460
Title: Cost Effective Air Filtration Intervention and Particulate Matter Monitoring in Low-Income Housing to Reduce Asthma Morbidity
Brief Title: Cost Effective Air Filtration Intervention in Low-Income Housing to Reduce Asthma Morbidity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Little Sisters of the Assumption Family Health Service (Unknown)
Responsible Party: Principal Investigator, Matthew S. Perzanowski, Professor of Environmental Health Sciences, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV8505; NYHHU009624 (Other Grant/Funding Number: US Department of Housing and Urban Development)
Record Dates: First submitted 2025-08-07; First posted 2025-08-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Asthma Attack; Lung Function; Airway Inflammation
Keywords: asthma; air cleaner; particulate matter; pm2.5; lung function; airway inflammation; children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled for a one-year trial of a HEPA air cleaner. All subjects will receive the air cleaner. Subjects will serve as their own controls. Given the existing evidence that air cleaners can reduce asthma morbidity, a sham or control group does not seem to be necessary nor ethically sound for this intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Air Cleaner Intervention (Experimental): Participants in this single arm of the study will be enrolled for a one-year trial of a HEPA air cleaner. Subjects will serve as their own controls.
  Interventions: Device: Austin Air Cleaner

INTERVENTIONS:
Device: Austin Air Cleaner — The Austin Air Purifier consists of 4 stages, a large particle pre-filter, medium pre-filter, a medical grade HEPA filter and a high efficiency gas arrestance carbon cloth to reduce air pollution in homes.

SUMMARY:
This project will investigate the effectiveness of HEPA air cleaners in reducing indoor air pollution and improving asthma morbidity in children living in East Harlem, New York City (NYC). The study will be conducted over a 2-year period.

Columbia University and Little Sisters of the Assumption Family Health Service (LSAFHS) will conduct an intervention study to evaluate the efficacy of using a cost-effective high-capacity high efficiency particulate air (HEPA) filter air cleaner to reduce airborne particulate matter (PM) in the homes of children with asthma and to reduce their asthma morbidity. The study will take place in East Harlem, a low-income neighborhood with high asthma prevalence. It will build on findings from prior Housing and Urban Development Lead and Healthy Homes Technical Studies (HUD LHHTS)-funded research, the experience of LSAFHS installing air cleaners in the homes of asthmatic children, and recent findings demonstrating the effectiveness of home air cleaners in reducing asthma morbidity. The investigators hypothesize that the cost-effective single air cleaner will substantially reduce PM exposure in the homes of asthmatic children and reduce airway inflammation and asthma morbidity. This study will use cutting-edge air sampling technology to continuously quantify and characterize indoor air pollutants in the home for one year, verify and incentivize compliance, and conduct repeated exhaled nitric oxide and pulmonary function tests before and throughout the year after the intervention. This cost-effective intervention can be easily and quickly implemented in homes in low-income, urban communities and easily transferred between homes if families move.

DETAILED DESCRIPTION:
The investigators propose an intervention study to evaluate if using a cost-effective high-capacity air filter will reduce air pollutants in the homes of asthmatic children and reduce their asthma symptoms. The study will take place in New York City, including East Harlem, a low-income, primarily Latino neighborhood with high asthma prevalence. The investigators hypothesize that a cost-effective single air cleaner placed in the homes of asthmatic children will substantially reduce air pollutants exposure and reduce airway inflammation and asthma symptoms. During the intervention, the study team will continuously monitor indoor air pollution by measuring particulate matter (tiny particles suspended in the air) for one year, verify and incentivize compliance, and conduct two types of breathing tests on the asthmatic child throughout the intervention: 1. One test measures exhaled nitric oxide (a gas collected by blowing air in a portable device, the levels of this gas are higher when there is inflammation in the airways), and 2. The second breathing test is a pulmonary function test (to measure lung capacity and diameter of the airways). The study team will also collect asthma symptom information through questionnaires. If successful, this study will provide evidence for a cost-effective intervention implemented without structural housing changes that can be easily and quickly implemented in homes in low-income urban communities. This study design will utilize a set of air monitors that will allow for high resolution quantification and characterization of particulate matter in the home before the intervention and one-year after placement of the air filter, which will allow researchers to better understand the impact of the filter on home air quality throughout the year. The study team will test the hypothesis that the single filter will substantially reduce particulate matter in the homes of asthmatic children and reduce airway inflammation and asthma morbidity in the child.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-18 years
* Asthma symptoms in the past 4 weeks
* Resident in lower-income housing in NYC Northern Manhattan and South Bronx

Exclusion Criteria:

* Inability to successfully perform spirometry maneuver or FeNO test
* Family planning to move in the next year

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Fractional Exhaled Nitric Oxide (FeNO) | 1 week before, immediately before, two weeks after, and one year after the air cleaner is turned on.
  A portable fractional exhaled nitric oxide (FeNO) monitor will used to measure exhaled NO, a biomarker of airway inflammation. FeNO will be measured at four timepoints with respect to the time the air cleaner is turned on.
Forced Expiratory Volume in 1 Second/ Forced Vital Capacity (FEV1/FVC) Ratio | 1 week before, immediately before, two weeks after, then once a month (up to 1 year) after the air cleaner is turned on.
  Easy to use, pocket-size spirometers (MIR) will be delivered to the homes along with the initial delivery of equipment. Subjects will be thoroughly trained on how to perform a pulmonary function test (PFT). These spirometers connect via Bluetooth to an application previously installed on the subject's cell phone. PFT data will be downloaded onto Columbia University computers from the app and the results will be scored and validated by trained personnel under the supervision of a spirometry expert.
  FEV1/FVC measures the proportion of vital capacity expired in the first second of forced expiration to the full forced vital capacity (how much air can be exhaled). FEV1/FVC will be measured at 15 timepoints with respect to the time the air cleaner is turned on.
Number of Attacks of Wheezing | Once per month for up to 12 months after the air cleaner is turned on
  The number of attacks of wheezing in the past 4 weeks will be reported.
Number of Emergency Department (ED) Visits | 12 months after the air cleaner is turned on
  Number of ED visits in the past year.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S Perzanowski, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared when the study results are published.
Supporting Information: Study Protocol, SAP
Time Frame: Shared data generated from this project will be made available as soon as possible, and no later than the time of publication or the end of the funding period, whichever comes first. The duration of preservation and sharing of the data will be a minimum of 10 years after the end of the funding period.
Access Criteria: All dataset(s) that can be shared will be deposited in the Data Archive for Demography and Population Sciences (DSDR). This repository is supported by the Inter-university Consortium for Political and Social Research (ICPSR).